CLINICAL TRIAL: NCT01606852
Title: Testing the Feasibility of Patient Controlled Sedation for Ventilated ICU Patients
Acronym: PCS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IND 111693; R21NR012795 (NIH)
Record Dates: First submitted 2012-04-09; First posted 2012-05-28 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Acute Respiratory Failure; Anxiety
Keywords: sedation; mechanical ventilation; anxiety; respiratory failure
MeSH Terms: conditions — Anxiety Disorders; Respiratory Insufficiency | interventions — Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- usual sedative practice (No Intervention): Subjects will have "usual care" sedation directed by their patient care team with no protocolized restriction on drug doses, selection or duration.
- Patient controlled sedation (Experimental): Subjects will be given the hand actuator connected to a Lifecare PCA Infusion System in the PCA + continuous mode with the syringe filled with 4 ucg/ml of dexmedetomidine. A loading dose (0.5 mcg/kg) will be given followed by a continuous basal infusion (0.2-0.7 mcg/kg/hr) with 3 allowable patient-controlled self-boluses per hour (0.25 mcg/kg) each with a 20-minute lock-out. Bedside RNs will adjust the basal rate to a maximum of based on the number of bolus requests in the prior two hours. Subjects can also receive bolus supplemental sedative medications (benzodiazepines and/or opioids)if needed in the judgment of the patient-care nurse.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — loading dose (0.5 mcg/kg i.v.), followed by a continuous basal infusion (0.2-0.7 mcg/kg/hr) with 3 allowable patient-controlled self-boluses per hour (0.25 mcg/kg) each with a 20-minute lock-out. Study infusion up to 5 days.
  Other Names: Administered via a Lifecare PCA Infusion System (Hospira)
  Arms: Patient controlled sedation

SUMMARY:
Mechanical ventilation (MV) is the most frequently used life-support modality in intensive care units (ICUs). To reduce anxiety, stress and promote tolerance of MV, nurses frequently administer a variety of sedative medications to their patients based on subjective observations.

The investigators hypothesize that patient-controlled sedation, compared to clinician-directed sedation, will decrease sedative exposure while decreasing patient anxiety during the episode of mechanical ventilation.

DETAILED DESCRIPTION:
A study to determine whether critically ill patients, during a substantial portion of their time on mechanical ventilation, can reduce anxiety symptoms better with PCS than their caregivers while reducing over-sedation, duration of mechanical ventilation and length of ICU stay will require hundreds of subjects enrolled on a multi-day protocol. However, patient-controlled sedation has been used in less than 20 patients and only for less than 24 hours. Therefore this study is designed to:

1. Establish the feasibility of subject recruitment and protocol adherence in a randomized pilot trial that compares patient-controlled sedation (PCS) using dexmedetomidine to usual sedation practice in mechanically ventilated patients. Feasibility will be defined by: a) number and proportion of patients or proxies who consent to enrollment, b) proportion of eligible subjects enrolled on Days 1,2,3,4 etc, of mechanical ventilation, c) number of days on protocol, up to five days, that subjects successfully use the PCS device, d) ability of ICU nurses to adjust the pump and adhere to the infusion rates of the PCS protocol.
2. Develop and refine the study protocol including: a) improving the proportion of patient daily assessments actually completed such as anxiety and delirium scales, b) develop a protocol to reliably determine when the subject is not able to self-manage their sedation due to weakness, confusion or severe illness; c) create rules for suspending PCS therapy and d) develop a post-ICU symptom interview.
3. Estimate effect sizes on key variables to inform the design of a future randomized trial to compare: a) sedative exposure, anxiety levels, and delirium occurrence between groups, b) adverse event rates and protocol violations related to the drug, pump or both; and c) duration of mechanical ventilation and ICU stay.

ELIGIBILITY:
Inclusion Criteria:

* adult intubated patients with respiratory failure expected to require mechanical ventilation for at least an additional 48 hours
* subjects have to have at least a 50% chance of being able to operate the PCS machine (i.e., adequate hand strength and cognition)

Exclusion Criteria:

* aggressive ventilatory support such as positive end expiratory pressure > 15 cm of water, prone ventilation, use of high-frequency oscillator ventilator
* hypotension requiring vasopressors (systolic blood pressure < 85 mmHg), second or third degree heart block or bradycardia (heart rate < 50 beats/min.)
* permanent condition preventing the use of push button device (e.g., paralysis)
* pregnancy or lactation
* acute hepatitis or liver failure
* general anesthesia 24 hours prior
* acute stroke or uncontrolled seizures
* acute MI
* severe cognition or communication problems (e.g., coma as main reason for intubation, deafness without signing literacy, dementia or severe delirium)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Craig Weinert, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Sedative Practice | Patient Controlled Sedation
Started | 7 | 8
Completed | 7 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Sedative Practice | Patient Controlled Sedation | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.5 (13.2) | 66.5 (13.2) | 66.5 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 6 | 7
  Male | 6 | 2 | 8
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Aggregate Sedative Exposure During PCS Use (up to 5 Days).
Description: Will use the sedation intensity score Scale is based on a score of 1 (full arousal) to 4 (no arousal)
Time Frame: 5 days after enrollment
Measure: Number (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Sedative Practice | Patient Controlled Sedation
Number analyzed (Participants) | 7 | 8
units on a scale | 4 [1 to 4] | 3.5 [1 to 4]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: arterial hypotension, bradycardia, self-extubations, and protocol violations related to drug, pump or both.
Time Frame: During 5 days of study protocol
Measure: Number; unit: participants
Arm/Group | Usual Sedative Practice | Patient Controlled Sedation
Number analyzed (Participants) | 7 | 8
participants | 7 | 8

ADVERSE EVENTS:
Arm/Group | Usual Sedative Practice | Patient Controlled Sedation
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 7/7 | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Sedative Practice (N=7) | Patient Controlled Sedation (N=8)
GI (Gastrointestinal disorders) | 5 (5) | 7 (7)
Heart (Cardiac disorders) | 1 (1) | 4 (4)
Skin (Infections and infestations) | 4 (4) | 4 (4)
Nervous System (Nervous system disorders) | 1 (1) | 2 (2)
Eye/Ear (General disorders) | 2 (2) | 0 (0)
Urinary (Renal and urinary disorders) | 2 (2) | 4 (4)
Sleep (General disorders) | 2 (2) | 3 (3)
Other (General disorders) | 3 (3) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No